CLINICAL TRIAL: NCT07094438
Title: Study Safety and Efficacy of Deep Brain Stimulation (DBS) and Cervical Deep Lymphoid-venous Anastomosis (LVA) in Patients With Severe Alzheimer's Disease
Brief Title: Study Safety and Efficacy of Deep Brain Stimulation (DBS) and Cervical Deep Lymphoid-venous Anastomosis (LVA) in Alzheimer's Disease
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Zhiqi Mao, Principal Investigator, Chinese PLA General Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: ChinaPLAGH_CNT
Record Dates: First submitted 2025-07-17; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DBS arm (Experimental): Patients in the DBS group underwent deep brain electrode implantation, followed by cranial MRI and CT to verify the accuracy of electrode placement.
  Interventions: Procedure: Deep Brain Stimulation, DBS
- LVA arm (Experimental): Patients in the LVA group underwent LVA surgery, followed by cervical ultrasound and CT to assess the anastomosis.
  Interventions: Procedure: Deep cervical lymphatic-venous anastomosis, LVA
- medication arm (Active Comparator): Patients in the medication group received drug therapy only, without undergoing surgery.
  Interventions: Drug: Recognized pharmacological treatments for AD.

INTERVENTIONS:
Procedure: Deep Brain Stimulation, DBS — Deep brain stimulation (DBS) is performed after preoperative MRI and CT images are fused in a planning system to determine the target and trajectory. Under general anesthesia, electrodes are precisely implanted into the fornix or nucleus basalis of Meynert using a stereotactic frame or neurosurgical robot. The electrodes are inserted through a burr hole in the patient's skull and connected to a pulse generator placed subcutaneously in the chest. Optimal stimulation parameters for Alzheimer's disease are not yet established. For fornix targets, settings are typically 3-3.5 V, ~130 Hz, 90 μs; for nucleus basalis targets, 2-4.5 V, 10-20 Hz, 90-150 μs, adjusted according to anatomical features and intraoperative responses.
  Arms: DBS arm
Procedure: Deep cervical lymphatic-venous anastomosis, LVA — Cervical deep lymphaticovenous anastomosis (LVA) microsurgically connects deep cervical lymphatic vessels to adjacent veins, promoting drainage of brain-derived amyloid-β and tau into the venous system and potentially alleviating Alzheimer's disease symptoms. The minimally invasive neck procedure involves small incisions and high-magnification suturing of lymphatics and veins with ultra-fine (11-0 or 12-0) sutures, creating multiple anastomoses to enhance brain lymphatic outflow.
  Arms: LVA arm
Drug: Recognized pharmacological treatments for AD. — Patients in the medication group received only the currently recognized pharmacological treatments for AD, including Memantine Hydrochloride and Donepezil.
  Arms: medication arm

SUMMARY:
To investigate the safety of deep brain stimulation (DBS) and cervical deep lymphoid-venous anastomosis (LVA) in the treatment of severe Alzheimer's disease (AD); to investigate the effectiveness of DBS and LVA in the treatment of severe AD, i.e., effects of deep brain stimulation on cognitive function, emotion and life quality in patients with severe AD.

ELIGIBILITY:
Inclusion Criteria:

* Meeting the diagnostic criteria for dementia formulated by the National Institute on Aging-Alzheimer's Association (NIA-AA).
* Clinical Dementia Rating (CDR) score of 3 points.
* Ability to ambulate independently or with the aid of a walker/cane.
* Adequate visual and auditory capacity to cooperate with examinations and treatment.
* Voluntary participation with written informed consent provided by both the subject and their legal guardian.

Exclusion Criteria:

* Pre-existing abnormal brain structure (e.g., tumor, cerebral infarction, hydrocephalus, or intracranial hemorrhage).
* Comorbidity with other neurological disorders such as multiple sclerosis, epilepsy, or Parkinson's disease.
* Psychiatric disorders: e.g., anxiety, depression, other affective disorders, or drug-induced psychosis.
* Severe internal diseases, currently using respiratory/cardiovascular/anticonvulsant/psychotropic drugs, or clinically significant gastrointestinal, renal, hepatic, respiratory, infectious, endocrine, or cardiovascular diseases, cancer, alcoholism, or substance addiction.
* Severe auditory or visual impairment.
* Clinical comorbidities with life expectancy <2 years.
* History of cranial surgery.
* Contraindications to MRI or transcranial alternating current stimulation (tACS) (e.g., cardiac pacemaker, post-deep brain stimulation surgery).
* Eczema or sensitive skin.
* Familial Alzheimer's disease.
* Other types of dementia: e.g., vascular dementia, Lewy body dementia, frontotemporal dementia, or infectious dementia;
* Any other condition deemed by the investigator as unsuitable for the study

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
The Alzheimer's Disease Assessment Scale cognitive subscale (ADAS-Cog) | changes of baseline and month 1, month 3, month 6, month 9, month 12, month 15, month 18 after surgery
  The Alzheimer's Disease Assessment Scale cognitive subscale (ADAS-Cog) scale is widely used for evaluating the severity of AD. ADAS-Cog consists of 12 components including word recall, naming, command, constructional praxis, ideational praxis, orientation, word recognition, remembering test instructions, spoken language ability, word finding difficulty, comprehension of oral language, and attention. The ADAS-Cog assesses multiple cognitive domains including memory, language, praxis, and orientation. ADAS-Cog score ranges from 0-75, with higher scores indicating more severe cognitive impairment.
Mini-Mental State Examination (MMSE) score | changes of baseline and month 1,month 3, month 6, month 9, month 12 month 15, month 18 after surgery
  Mini-Mental State Examination (MMSE) is one of the most influential cognitive screening tools worldwide. It consists of five dimensions including orientation (10 points), registration (3 points), attention and calculation (5 points), recall (3 points) and language and praxis (9 points). Educational attainment level-related dementia classification: illiterate: 5 points ≤ MMSE score ≤16 points; primary school: 8 points ≤ MMSE score ≤ 20 points; junior high school and above: 10 points ≤ MMSE score ≤ 24 points.
Clinical Dementia Rating(CDR) score | changes of baseline and month 1, month 3, month 6, month 9, month 12, month 15, month 18 after surgery
  The Clinical Dementia Rating(CDR) is 5-point scale used to characterize six domains (memory, orientation, judgment & problem solving, community affairs, home & hobbies and personal care) of the cognitive and functional performance of the aged (in particular AD patients). Patients are rated on dementia severity: 0 = normal, 0.5 = questionable dementia; 1 = mild dementia; 2 = moderate dementia; 3 = severe dementia.

CONTACTS AND LOCATIONS:
Overall Officials: Zhiqi Mao, Ph.D, Principal Investigator — Chinese PLA General Hospita
Locations (1):
- Chinese PLA General Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided